CLINICAL TRIAL: NCT01526967
Title: Observational Evaluation of the Peristomal Skin Condition in Ostomates Using ConvaTec Moldable Technology™ Skin Barriers
Brief Title: Observational Evaluation of the Peristomal Skin Condition in Ostomates
Acronym: OSMOSE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-0509-12-U359
Record Dates: First submitted 2012-02-01; First posted 2012-02-06 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Ostomy
Keywords: ostomy; peristomal skin breakdown; ConvaTec Moldable Skin Barriers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- New moldable user: Subjects presenting with peristomal lesions with a traditional barrier and for whom a ConvaTec Moldable Technology™ Skin Barrier is used as a replacement.
- New osomate: Subjects for whom a ConvaTec Moldable Technology™ Skin Barrier is used as the first long-term (within 7 days of ostomy surgery) system following surgery and have intact peristomal skin.

SUMMARY:
The purpose of this study is to estimate the incidence and severity of peristomal skin lesions and evaluate the progression of the peristomal skin condition at 8-15 days following application of the barrier.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 18 years old and older.
* Subjects who agree to participate in the evaluation and who have signed the informed consent form.
* Subjects presenting with a stoma (ileostomy, colostomy or urostomy).
* Subjects for whom a ConvaTec Moldable Technology™ Skin Barrier per package insert is used as the first long-term (within 7 days of ostomy surgery) system following surgery and have intact peristomal skin.

OR

* Subjects presenting with peristomal skin lesions using a traditional barrier and for whom a decision to replace the traditional barrier with ConvaTec Moldable Technology™ Skin Barrier per package insert is made in the context of routine clinical care.

Exclusion Criteria:

* Subjects who, according to the investigator, have cognitive problems that prevent them from answering a questionnaire or for whom the evaluation could be a problem.
* Subjects who are in a simultaneous clinical evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colostomates, ileostomates, urostomates in acute care settings or community at large.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Peristomal skin condition | At day 12
  Change in peristomal skin condition from baseline as assessed with the SACS Instrument

SECONDARY OUTCOMES:
Peristomal skin condition | at 1 month
  Change in peristomal skin condition from baseline as assessed with the SACS instrument
Level of satisfaction | At 2 months
  Subjects satisfaction as measured with a satisfaction survey
Accessory usage | Up to 2 months
  Subjects use of additional products in stoma care.
Peristomal Skin Condition | At 2 months
  Change in peristomal skin condition from baseline as assessed with the SACS instrument
Level of satisfaction | At 12 days
  Subjects level of satisfaction as measured by a satisfaction survey
Level of satisfaction | At 1 month
  Subjects level of satisfaction as measured with a satisfaction survey

CONTACTS AND LOCATIONS:
Overall Officials: Qing Li, Ph.D, MD, Study Chair — ConvaTec Inc.
Locations (13):
- United States (13):
  - Independent Nurse Consultant, Tucson, Arizona
  - John Muir Health Concord Campus, Concord, California
  - Conn. Clinical Nursing Associate, LLC, Plymoth, Connecticut
  - Baptist Home Health, Jacksonville, Florida
  - Porter Hospital, Valparaiso, Indiana
  - Serena Group - Dr. Thomas Serena MD, Cambridge, Massachusetts
  - Henry Ford Macomb Hospital, Clinton Township, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - St. Anthony's Medical Center, St Louis, Missouri
  - ID Med Inc., Columbus, Ohio
  - RI Colorectal Clinic, LLC, Pawtucket, Rhode Island
  - San Jacinto Methodist Hospital, Baytown, Texas
  - NW Pavillion Ostomy Clinic, Renton, Washington